CLINICAL TRIAL: NCT01673269
Title: Prospective Study of the Risk of Bacteremia in Directed Cholangioscopic Examination of the CBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Collaborators: American College of Gastroenterology (Other)
Responsible Party: Principal Investigator, Mohamed O Othman, Assistant Professor, Texas Tech University Health Sciences Center, El Paso
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: E12053-A
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Choledocholithiasis; Cholangiocarcinoma; Benign Stricture of Common Bile Duct
Keywords: ERCP; Direct cholangioscopic examination of the common bile duct; Choledocholithiasis; Cholangiocarcinoma; Benign stricture of common bile duct
MeSH Terms: conditions — Choledocholithiasis; Cholangiocarcinoma | interventions — Blood Culture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ERCP with direct examination of the CBD (Experimental)
  Interventions: Other: Blood culture ( aerobic and anaerobic)

INTERVENTIONS:
Other: Blood culture ( aerobic and anaerobic) — Blood culture 5 minutes and 30 minutes after the procedure

SUMMARY:
When a doctor performs Endoscopic retrograde cholangiopancreatography "ERCP" (Endoscopy to examine the bile duct) a flexible tube is inserted into the mouth and into the stomach. The tube passes beyond the stomach and into an opening in the liver called the bile duct. Another small flexible endoscope is inserted inside the ERCP scope to directly visualize the bile duct to ensure that there are no cancers or stones in the bile duct and occasionally to take a sample from the bile duct. The purpose of our study is to examine wither performing this procedure can transmit bacteria from the bile duct to the main blood stream.

DETAILED DESCRIPTION:
This is a prospective study to measure the frequency of bacteremia in patients undergoing ERCP with direct cholangioscopic examination of the Common Bile Duct "CBD". A blood culture will be drawn from patients prior to the procedure, 5 minutes after the procedure and 30 minutes after the procedure. The patient will be followed up for 7 days after procedure for fever and sepsis. The estimated sample size is 60 patients.

ELIGIBILITY:
Inclusion Criteria:

* 1- Adult patients (18-80) who are undergoing ERCP with direct cholangioscopic examination of the common bile duct to ensure the clearance of the common bile duct from stones.

  2- Adult patients (18-80) who are undergoing ERCP with direct cholangioscopic examination of the common bile duct for stone removal.

  3- Adult patients (18-80) who are undergoing ERCP with direct cholangioscopic examination of the common bile duct for tissue acquisition from the common bile duct mass.

  4- Adult patients (18-80) who are undergoing ERCP with direct cholangioscopic examination of the common bile duct for tissue acquisition from common bile duct strictures.

Exclusion Criteria:

* 1- Patients younger than 18 yrs old or older than 80 yrs. 2- Pregnant patients. 3- Patient with ascending cholangitis, pneumonia or urinary tract infection 4- Patients who received antibiotics in the last 2 weeks prior to the procedure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
the frequency of bacteremia after ERCP with direct cholangioscopic examination of the CBD | 5 minutes and 30 minutes
  To measure the frequency of bacteremia after ERCP with direct cholangioscopic examination of the CBD by obtaining blood culture 5 minutes and 30 minutes after the procedure

SECONDARY OUTCOMES:
To measure the frequency of fever or sepsis after ERCP with direct cholangioscopic examination of the CBD | within 24 hours and one week of the procedures.
  This outcome will be obtained by calling the patient 24 hour and 1 week after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed O Othman, MD, Principal Investigator — Texas Tech University at El Paso
Locations (1):
- Texas Tech University Health Sciences Center at El Paso, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Othman MO, Guerrero R, Elhanafi S, Davis B, Hernandez J, Houle J, Mallawaarachchi I, Dwivedi AK, Zuckerman MJ. A prospective study of the risk of bacteremia in directed cholangioscopic examination of the common bile duct. Gastrointest Endosc. 2016 Jan;83(1):151-7. doi: 10.1016/j.gie.2015.05.018. Epub 2015 Jun 23. PMID 26116469